CLINICAL TRIAL: NCT01039441
Title: The Effect of Local Anesthesia and Simple Maneuver on Shoulder Pain After Gynecologic Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Duk Soo Bae/Chairman of Dept. of Ob. & Gyn, The department of obstetrics and gynecology, Samsung Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-07-071
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Last update posted 2009-12-25 (Estimated); Status verified 2008-10

CONDITIONS: Gynecologic Laparoscopic Surgery for Benign Adnexa Disease
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- instillation of normal saline 50ml under the diaphragm (Placebo Comparator)
  Interventions: Other: normal saline
- the instillation of 0.5% bupivacaine under the diaphragm (Experimental)
  Interventions: Procedure: Intraperitoneal instillation of bupivacaine
- CO2 removal by means of a pulmonary recruitment maneuver (Experimental)
  Interventions: Procedure: CO2 removal by means of a pulmonary recruitment maneuver
- the instillation of bupivacaine + CO2 removal by maneuver (Experimental)
  Interventions: Procedure: Intraperitoneal instillation of bupivacaine +CO2 removal by means of a pulmonary recruitment maneuver

INTERVENTIONS:
Procedure: Intraperitoneal instillation of bupivacaine — A mixture of 50ml solution (20ml of 0.5% bupivacaine + 30ml normal saline) is instilled under the diaphragm.
  Arms: the instillation of 0.5% bupivacaine under the diaphragm
Procedure: CO2 removal by means of a pulmonary recruitment maneuver — CO2 is removed by means of a pulmonary recruitment maneuver consisting of five manual inflations of the lung with a maximum pressure of 30 cm H2O
  Arms: CO2 removal by means of a pulmonary recruitment maneuver
Procedure: Intraperitoneal instillation of bupivacaine +CO2 removal by means of a pulmonary recruitment maneuver
  Arms: the instillation of bupivacaine + CO2 removal by maneuver
Other: normal saline
  Arms: instillation of normal saline 50ml under the diaphragm

SUMMARY:
This prospective, randomized controlled trial was designed to compare the efficacy of a simple maneuver using lower airway pressure (30 cm H2O) and intraperitoneal instillation of bupivacaine, alone or in combination, to reduce shoulder pain after gynecologic laparoscopy.

Patient aged 15-65 years, scheduled for laparoscopic surgery for benign adnexa disease will be eligible for the study. Patients will be excluded from analysis if the procedure requires conversion to a laparotomy, an operative time > 3 hours, or interpretation of pain is impossible due to serious adverse effects

240 patients will be randomly assigned to one of four groups Upon completion of surgery, the patient is placed in the Trendelenburg position (30 degrees), and one of four procedures is followed. For group A (control), 50 ml of normal saline is instilled under the diaphragm and CO2 is removed by manual deflation of the abdominal cavity through the cannula; For group B, a mixture of 50ml solution (20ml of 0.5% bupivacaine + 30ml normal saline) is instilled under the diaphragm and CO2 is removed by manual deflation of the abdominal cavity through the cannula; For group C, 50 ml of normal saline is instilled under diaphragm and CO2 was removed by means of a pulmonary recruitment maneuver consisting of five manual inflations of the lung with a maximum pressure of 30 cm H2O. The anesthesiologist holds the fifth positive pressure inflation for approximately 5 seconds. During these maneuvers, the surgeon will be instructed to ensure that the trocar sleeve valve is fully open to allow the CO2 gas to escape. For group D, patients receive an instillation of a mixture of 50ml solution in combination with the clinical maneuver.

Patients will be given a questionnaire with the pain question represented as a visual analog scale (VAS) preoperatively. Patients will be asked to fill out the questionnaires during the first 24 hours after surgery to determine the frequency and severity of their shoulder pain. All patients are instructed to record the pain scores regarding their shoulder pain only. The degree of postoperative shoulder pain will be assessed using VAS at 1, 6, 12, and 24 hours postoperatively. The VAS, with scores ranging from 0 (no pain) to 10 (excruciating pain), is constructed without numeration, thus allowing patients to mark a point along the scale that best represented their pain at that time.

In addition, the following parameters are recorded on the case report form by the investigators: operative time, blood loss, the length of hospital stay, analgesic use, and incidence of postoperative events.

ELIGIBILITY:
Inclusion Criteria:

* benign adnexa diseases which are scheduled for laparoscopic surgery

Exclusion Criteria:

* The procedure required conversion to a laparotomy, An operative time > 3 hours, Interpretation of pain was impossible due to serious adverse effects.

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The degree of shoulder pain after gynecologic laparoscopy | During the first 24hours after surgery; 1,6, 12, 24hr

CONTACTS AND LOCATIONS:
Overall Officials: Duk Soo Bae, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho M, Kim CJ, Hahm TS, Lee YY, Kim TJ, Lee JW, Kim BG, Bae DS, Choi CH. Combination of a pulmonary recruitment maneuver and intraperitoneal bupivacaine for the reduction of postoperative shoulder pain in gynecologic laparoscopy: a randomized, controlled trial. Obstet Gynecol Sci. 2020 Mar;63(2):187-194. doi: 10.5468/ogs.2020.63.2.187. Epub 2020 Feb 20. PMID 32206659